CLINICAL TRIAL: NCT00984867
Title: A 24-week, Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, International Phase III Study With 24 Week Extension to Evaluate the Safety and Efficacy of Dapagliflozin 10 mg/Day in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control on a DPP-4 Inhibitor Sitagliptin+/-Metformin
Brief Title: Dapagliflozin DPPIV Inhibitor add-on Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00010
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes
Keywords: Dapagliflozin DPP IV inhibitor add on study; Inadequate control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Dapagliflozin 10 mg tablet
  Interventions: Drug: Dapagliflozin
- 2 (Placebo Comparator): Matching placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg tablet, oral, once daily, 48 weeks
  Arms: 1
Drug: Placebo — Matching placebo tablet
  Arms: 2

SUMMARY:
This study aims to investigate how dapagliflozin can control blood sugar in patients with type 2 diabetes when added to existing treatments (sitagliptin alone or in combination with metformin). The effect of dapagliflozin on weight and blood pressure will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Patients who are not receiving treatment , or those who currently receive metformin, sitagliptin or vildagliptin or the combination of these
* Patients will be screened by a blood test and only those who need additional therapy can be enrolled

Exclusion Criteria:

* Patients with type 1 diabetes
* Patients with very poorly controlled diabetes
* Any clinically significant illness, which in the judgement of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Jabbour, MD, Principal Investigator — Thomas Jefferson University, Philadelphia
Locations (88):
- United States (45):
  - Research Site, Huntsville, Alabama
  - Research Site, Ozark, Alabama
  - Research Site, Anaheim, California
  - Research Site, Chula Vista, California
  - Research Site, Greenbrae, California
  - Research Site, Laguna Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Riverside, California
  - Research Site, West Hills, California
  - Research Site, Boca Raton, Florida
  - Research Site, DeLand, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Longwood, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Orange, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Stone Mountain, Georgia
  - Research Site, Wichita, Kansas
  - Research Site, Lake Charles, Louisiana
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Pahrump, Nevada
  - Research Site, Staten Island, New York
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medord, Oregon
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Simpsonville, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, North Richland Hills, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burke, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Lakewood, Washington
- Argentina (10):
  - Research Site, Berazategui, Buenos Aires
  - Research Site, La Plata, Buenos Aires
  - Research Site, Lanús, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Morón, Buenos Aires
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Caba, Buenos Aires F.D.
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Salta, Salta Province
  - Research Site, Santa Fe, Santa Fe Province
- Germany (8):
  - Research Site, Bad Nauheim
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Hamburg
  - Research Site, Meissen
  - Research Site, Münster
  - Research Site, Pirna
  - Research Site, Wangen
- Mexico (2):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
- Poland (12):
  - Research Site, Ciechocinek
  - Research Site, Czechowice-Dziedzice
  - Research Site, Gdansk
  - Research Site, Gniewkowo
  - Research Site, Krakow
  - Research Site, Krotoszyn
  - Research Site, Mrągowo
  - Research Site, Poznan
  - Research Site, Sopot
  - Research Site, Torun
  - Research Site, Zabrze
  - Research Site, Łęczyca
- United Kingdom (11):
  - Research Site, Bolton, Lancs
  - Research Site, Burbage, Leicester
  - Research Site, Sunbury-on-Thames, Middlesex
  - Research Site, Wansford, Peterborough
  - Research Site, Ecclesfield, Sheffield
  - Research Site, Addlestone, Surrey
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Coventry
  - Research Site, Harrow

REFERENCES:
- [Result] Jabbour SA, Hardy E, Sugg J, Parikh S; Study 10 Group. Dapagliflozin is effective as add-on therapy to sitagliptin with or without metformin: a 24-week, multicenter, randomized, double-blind, placebo-controlled study. Diabetes Care. 2014;37(3):740-50. doi: 10.2337/dc13-0467. Epub 2013 Oct 21. PMID 24144654
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- See also: D1690C00010_Clinical_Study_Report_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=292&filename=D1690C00010_Study_Synopsis_1Mar2012.pdf
- See also: D1690C00010_Revised_CSP1_and_Amdt_1_Priv_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=292&filename=D1690C00010_Revised_CSP1_and_Amdt_1_Priv_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 10 Oct 2009. Last participant last visit for 24-week period: 10 Mar 2011. 833 participants were enrolled, 452 randomized and 451 treated in 3 European countries, USA, Argentina and Mexico. Participants with T2DM who showed inadequate glycemic control (7.0% ≤ HbA1c ≤ 10.0% at randomization) on sitagliptin +/- metformin.
Pre-assignment Details: During a placebo lead-in period, participants were counselled on dietary and life-style modifications. Participants eligible for the study were stratified according to use of metformin.
Groups:
- Placebo: Placebo plus sitagliptin alone or in combination with metformin
- Dapagliflozin: Dapagliflozin 10 mg plus sitagliptin alone or in combination with metformin
Period: Overall Study
Arm/Group | Placebo | Dapagliflozin
Started | 226 (Of the 226 randomized and treated participants only 224 were included in the full analysis set.) | 225 (Of the 225 randomized and treated participants only 223 were included in the full analysis set.)
Completed | 203 | 208
Not Completed | 23 | 17
Not completed — Adverse Event | 3 | 7
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Lost to Follow-up | 3 | 4
Not completed — Poor/non-compliance | 0 | 1
Not completed — Subject no longer meets study criteria | 1 | 1
Not completed — site closing | 1 | 0
Not completed — lack of efficacy and subject compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapagliflozin | Total
Number analyzed (Participants) | 224 | 223 | 447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.0 (10.20) | 54.8 (10.42) | 54.9 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 96 | 202
  Male | 118 | 127 | 245
HbA1c [Mean (Standard Deviation); unit: HbA1c [%]] | 7.97 (0.778) | 7.90 (0.806) | 7.93 (0.792)
Body weight [Mean (Standard Deviation); unit: kg] | 89.23 (20.887) | 91.02 (21.637) | 90.12 (21.259)
FPG [Mean (Standard Deviation); unit: mg/dL] | 162.97 (34.452) | 162.19 (36.825) | 162.58 (35.618)
Seated SBP in subjects with baseline seated SBP ≥130 mmHg [Mean (Standard Deviation); unit: mmHg] | 139.30 (8.507) | 140.46 (8.018) | 139.85 (8.279)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To compare the change from baseline in HbA1c after 24 weeks treatment (LOCF) between dapagliflozin and placebo in patients with type 2 diabetes who are inadequately controlled on sitagliptin alone or on sitagliptin plus metformin.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 223 | 223
Percent | 0.04 (0.0509) [-0.06 to 0.14] | -0.45 (0.0509) [-0.55 to -0.35]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0. The study consisted of two strata: sitagliptin monotherapy group and sitagliptin plus metformin group; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.05 (2-sided). A hierarchical closed testing procedure was used to control Type I error across the primary & key secondary objectives, based on data from both strata combined; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.62 to -0.34], Standard Error of Mean 0.0720

2. Secondary Outcome: Adjusted Mean Change in Body Weight
Description: To compare the change in total body weight achieved with dapagliflozin versus placebo from baseline to week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Groups:
- Placebo: Placebo plus sitagliptin alone or in combination with metformin. Full analysis set.
- Dapagliflozin: Dapagliflozin 10 mg plus sitagliptin alone or in combination with metformin. Full analysis set.
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 224 | 223
kg | -0.26 (0.1741) [-0.60 to 0.09] | -2.14 (0.1745) [-2.48 to -1.80]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -1.89, 95% CI 2-sided [-2.37 to -1.40], Standard Error of Mean 0.2466

3. Secondary Outcome: Adjusted Mean Change in HbA1c in Participants With Baseline HbA1c ≥8%
Description: To compare the change in HbA1c in participants with baseline HbA1c ≥8% achieved with dapagliflozin versus placebo from baseline to week 24.
Time Frame: Baseline to Week 24
Population: Full analysis set, participants with baseline HbA1c >=8% and Week 24 (LOCF) value
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 99 | 94
Percent | 0.03 (0.0775) [-0.12 to 0.18] | -0.80 (0.0797) [-0.96 to -0.65]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.05 to -0.62], Standard Error of Mean 0.1106

4. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG)
Description: To compare the change in FPG achieved with dapagliflozin versus placebo from baseline to week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 222 | 222
mg/dL | 3.81 (2.3474) [-0.80 to 8.42] | -24.11 (2.3474) [-28.73 to -19.50]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -27.92, 95% CI 2-sided [-34.45 to -21.40], Standard Error of Mean 3.3200

5. Secondary Outcome: Adjusted Mean Change in Seated Systolic Blood Pressure (SBP) in Participants With Baseline SBP>=130 mmHg
Description: To compare the change in seated systolic blood pressure (SBP) in participants with baseline seated SBP >=130 achieved with dapagliflozin versus placebo from baseline to week 8.
Time Frame: Baseline to Week 8
Population: Full analysis set, participants with baseline SBP>=130mmHg and Week 8 (LOCF) value
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 111 | 101
mmHg | -5.12 (1.0211) [-7.14 to -3.11] | -5.98 (1.0638) [-8.08 to -3.89]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5583, ANCOVA — Not significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -0.86, 95% CI [-3.75 to 2.03], Standard Error of Mean 1.4659

6. Secondary Outcome: Adjusted Mean Change in 2-hour Post Liquid Meal Glucose Rise
Description: To compare the change in 2-hour post liquid meal glucose rise achieved with dapagliflozin versus placebo from baseline to week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 197 | 205
mg/dL | -6.84 (2.5098) [-11.77 to -1.90] | -21.65 (2.4604) [-26.49 to -16.81]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA — Not significant. Hierarchical testing procedure stopped at previous endpoint; with treatment group and stratum as effect and baseline value as covariate; Mean Difference (Final Values) = -14.82, 95% CI 2-sided [-21.73 to -7.90], Standard Error of Mean 3.5160

7. Secondary Outcome: Proportion of Participants Achieving a Therapeutic Glycemic Response Defined as a Reduction in HbA1c of ≥0.7% Compared to Baseline
Description: To compare the proportion of participants achieving a therapeutic glycaemic response, defined as a reduction in HbA1c of ≥0.7% compared to baseline, with dapagliflozin versus placebo at week 24. Least Squares Mean represents the percent of participants adjusted for HbA1c baseline value.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Dapagliflozin
Number analyzed (Participants) | 223 | 223
Percentage of participants | 16.6 (2.491) [11.7 to 21.4] | 35.3 (3.083) [29.3 to 41.2]
Statistical Analysis 1: Comparison: Placebo vs Dapagliflozin; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; Regression, Logistic — Not significant. Hierarchical testing procedure stopped at previous endpoint; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline value and stratum; Risk Difference (RD) = 18.7, 95% CI 2-sided [11.1 to 26.4], Standard Error of Mean 41.2

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment plus 4/30 days or up to follow-up visit if earlier, or up to and including the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Groups:
- Placebo: Placebo plus sitagliptin alone or in combination with metformin. Safety analysis set.
- Dapagliflozin: Dapagliflozin 10 mg plus sitagliptin alone or in combination with metformin. Safety analysis set.
Arm/Group | Placebo | Dapagliflozin
Serious Adverse Events (participants affected / at risk) | 9/226 | 10/225
Other Adverse Events (participants affected / at risk) | 14/226 | 9/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=226) | Dapagliflozin (N=225)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Medical device pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=226) | Dapagliflozin (N=225)
Nasopharyngitis (Infections and infestations) | 14 | 9

LIMITATIONS AND CAVEATS:
For participants who did not complete 8 and/or 24 weeks, respectively, LOCF was used. All endpoints were evaluated by excluding data after rescue with the exception of systolic blood pressure which was evaluated regardless of rescue medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.